CLINICAL TRIAL: NCT00298194
Title: The Effects of Z-338 on the Symptomatic Response to a Nutrient Challenge and Gastric Nutrient Distribution and Emptying in Subjects With and Without Functional Dyspepsia
Brief Title: The Effects of Z-338 in Subjects With and Without Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 99010205E
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Z 338

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Z-338

SUMMARY:
To assess in subjects with and without functional dyspepsia the effects of Z-338 on:

1. Type and severity of symptoms a standardized nutrient challenge
2. The gastric nutrient distribution and gastric emptying of a standardized nutrient challenge
3. The association of the above with the manifestations of symptoms and symptom pattern

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with functional dyspepsia Positive documented diagnosis of FD via RomeII criteria and three or more moderate symptoms of Gastrointestinal Score
2. Subjects with no history of functional dyspepsia Clinical assessment, physical examination and laboratory testing without evidence for relevant abnormality.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Holtmann, Professor, Principal Investigator — Royal Adelaide Hospital
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia